CLINICAL TRIAL: NCT03097978
Title: Clinical Trials of Pattern Recognition, Electrode Grid, RIC Arm in TMR Subjects
Brief Title: Comparison of Pattern Recognition Control and Direct Control in TMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Todd Kuiken, Director, Center for Bionic Medicine, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Single Group | Purpose: Basic Science
Other Study IDs: STU00068547
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Amputation; Amputation; Traumatic, Arm, Upper

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- RIC arm system with pattern recognition (Experimental): Subject will be fit with a custom socket and receive training on pattern recognition with the RIC arm prosthesis. Once appropriate training has occurred, outcome measures will be completed followed by a home trial for at least 6 weeks with the device. Outcome measures will be collected at the conclusion of the 6 week home trial.
  Interventions: Device: RIC arm system; Other: Pattern Recognition
- RIC arm system with direct control (Experimental): Subject will be fit with a custom socket and receive training on direct control with the RIC arm prosthesis. Once appropriate training has occurred, outcome measures will be completed followed by a home trial for at least 6 weeks with the device. Outcome measures will be collected at the conclusion of the 6 week home trial.
  Interventions: Device: RIC arm system; Other: Direct Control
- Commercial system with PR control (Experimental): Subject will be fit with a custom socket and receive training on pattern recognition with a conventional, commercial prosthesis system. Once appropriate training has occurred, outcome measures will be completed followed by a home trial for at least 6 weeks with the device. Outcome measures will be collected at the conclusion of the 6 week home trial.
  Interventions: Device: Commercial system; Other: Pattern Recognition
- Commercial system with Direct Control (Experimental): Subject will be fit with a custom socket and receive training on direct control with a conventional, commercial prosthesis system. Once appropriate training has occurred, outcome measures will be completed followed by a home trial for at least 6 weeks with the device. Outcome measures will be collected at the conclusion of the 6 week home trial.
  Interventions: Device: Commercial system; Other: Direct Control

INTERVENTIONS:
Device: Commercial system — Transhumeral amputees who have had TMR will use a commercially available prosthesis with an elbow,wrist, and a hand with custom electronics and software for both direct and pattern recognition - based control.
  Arms: Commercial system with Direct Control; Commercial system with PR control
Device: RIC arm system — Transhumeral amputees who have had TMR will use the RIC arm system prosthesis with an elbow,wrist, and a hand with custom electronics and software for both direct and pattern recognition - based control.
  Arms: RIC arm system with direct control; RIC arm system with pattern recognition
Other: Direct Control — Transhumeral amputees who have had TMR will use either a commercially available prosthesis or the RIC arm system prosthesis with an elbow,wrist, and a hand with custom electronics and software for both direct control.
  Arms: Commercial system with Direct Control; RIC arm system with direct control
Other: Pattern Recognition — Transhumeral amputees who have had TMR will use either a commercially available prosthesis or the RIC arm system prosthesis with an elbow,wrist, and a hand with custom electronics and software for pattern recognition control.
  Arms: Commercial system with PR control; RIC arm system with pattern recognition

SUMMARY:
Targeted Muscle Reinnervation increases the control signals available for commercial arm systems. A new type of control, pattern recognition, has been developed into a form that allows use with commercially available arm system. The goal of this project is a home trial, in which people who have had TMR will try the new controls and the new arm to find out if they are better than what is currently available. Home trials will also allow us to see what needs to be done to make our inventions work even better.

DETAILED DESCRIPTION:
Subjects who participate return to RIC several times (approximately 6-8 times) to undergo any necessary training and testing. Each visit will last from 2-5 days. The study will include use of up to three different prosthesis control systems at home for approximately 6 weeks each. The order of the systems will be randomized.

The first visit will allow us to cast the subject's residual limb for a socket and measure for a gel liner to be made with embedded electrode contacts prior to the next return. The socket interface will be fit for optimal comfort and a suspension sleeve and/or other straps, fasters, etc to best hold the prosthesis securely on the residual limb for the activities required. Unless changes are needed due to changes in limb volume, the same socket can be used for all phases of the study. During the initial and subsequent visits, subjects may practice the various control methods using a virtual reality system. EMG data and virtual "games" will be used to practice the control and will provide quantitative data that can be used to assess the various control methods mathematically, without the prosthesis.

Each phase of the study (up to 4 phases), will include preliminary training and testing at RIC lasting for 1-5 days, followed by approximately 6 weeks of at-home use of the system. After this time subjects will return to the RIC for 2-3 days of testing. They will then be trained and pre-tested in use of the next control during the same visit or at a later date. These systems include a commercially available myoelectric prosthesis with standard control, a commercially available device with advanced control (called pattern recognition), a commercially available device with pattern recognition and a new electrode configuration. Photographs or video recordings will be made during participation in this research study. These pictures and video recordings are essential for proper data analysis.

During the at-home use periods subjects will go about their daily business using the test prosthesis and will be asked document the experience with the prosthesis via weekly phone communication with study staff. Dates/times will be coordinated during normal business hours At the end of the at-home use period subjects will return to RIC for 3-5 days, where they will be asked to complete a questionnaire about how the prosthesis worked, and will undergo some non-invasive testing to see how well they can control and use the prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* A upper limb amputation at the transhumeral or shoulder-disarticulation level
* Successful TMR surgery
* Previous success at operating a myoelectric prosthesis using surface EMG signals from reinnervated muscles (not necessarily current prosthesis usage, although current prosthesis users may be more likely to use their trial prostheses).

Exclusion Criteria:

* Significant new injury that would prevent use of a prosthesis: The ability to consistently wear a prosthesis and perform activities of daily living and specific performance tasks is necessary to evaluate the relative benefits of the interventions.
* Cognitive impairment sufficient to adversely affect understanding of or compliance with study requirements, ability to communicate experiences, or ability to give informed consent: The ability to understand and comply with requirements of the study is essential in order for the study to generate useable, reliable data. The ability to obtain relevant user feedback through questionnaires and informal discussion adds significant value to this study. Of note, all TMR patients to date have normal cognitive function and we are not aware of any new brain injuries that would preclude participation
* Significant other co morbidity: Any other medical issues or injuries that would preclude completion of the study, use of the prostheses, or that would otherwise prevent acquisition of useable data by researchers.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Pattern recognition and the RIC arm system will demonstrate a significant improvement over exiting technology. | 15 months from initial enrollment
  Improved control of prosthesis as seen through functional use improvements.

SECONDARY OUTCOMES:
Modified Box and Blocks | At 1 month, 2 months, 4 months, 6 months
  Timed task to assess prosthetic control.
Jebsen Test of Hand Function | At 1 month, 2 months, 4 months, 6 months
  7 part timed diagnostic test to determine the level of hand function
Southampton Hand Assessment Procedure (SHAP) | At 1 month, 2 months, 4 months, 6 months
  The test consists of the manipulation of a series of both lightweight and heavyweight abstract objects. The procedure is designed to provide a score of functionality.
ACMC | At 1 month, 2 months, 4 months, 6 months
  Assessment of capacity for myoelectric prosthetic control

CONTACTS AND LOCATIONS:
Overall Officials: Todd Kuiken, MD, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hargrove L, Miller L, Turner K, Kuiken T. Control within a virtual environment is correlated to functional outcomes when using a physical prosthesis. J Neuroeng Rehabil. 2018 Sep 5;15(Suppl 1):60. doi: 10.1186/s12984-018-0402-y. PMID 30255800